CLINICAL TRIAL: NCT05299879
Title: Screening for Advanced Heart Failure IN Stable ouTpatientS (The SAINTS Study) - Early Identification of Advanced Heart Failure
Brief Title: Screening for Advanced Heart Failure IN Stable ouTpatientS - The SAINTS Study
Acronym: SAINTS-A
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Finn Gustafsson, Sponsor-Investigator, Rigshospitalet, Denmark
Other Study IDs: RH-SAINTS-A
Record Dates: First submitted 2022-03-07; First posted 2022-03-29 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Advanced heart failure; Screening
MeSH Terms: interventions — Exercise Test; Echocardiography; Walk Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Full blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symptomatic patients with HFrEF corresponding to NYHA II-III
  Interventions: Diagnostic Test: Cardiopulmonary exercise test, NT-proBNP, Echocardiography, 6 minute walk test, Right heart catheterization

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary exercise test, NT-proBNP, Echocardiography, 6 minute walk test, Right heart catheterization — Screening for advanced HF with modified criteria from the Heart Failure Association of the European Society of Cardiology

SUMMARY:
The purpose of the Screening for Advanced heart failure IN stable ouTpatientS (SAINTS) study is to determine the prevalence of advanced heart failure (HF) in symptomatic patients with HF and reduced left ventricular ejection fraction (HFrEF), corresponding to the New York Heart Association functional class II-III.

Recognition of advanced HF is a challenge for physicians and under referral for advanced management is a considerable problem. There are excellent treatment options for patients with advanced HF, i.e. heart transplantation or left ventricular assist device (LVAD) implantation, and outcomes with these therapies are considerably better if patients are treated before irreversible end-organ damage occurs. International consensus highlights the importance of timely recognition and referral of these patients to advanced HF centers.

The investigators aim to screen patients with symptomatic HFrEF who are followed in Danish HF clinics in the Copenhagen region with echocardiography, cardiopulmonary exercise test, 6 minute walk test, and NT-proBNP. The investigators hypothesize that 20% of patients with symptomatic heart failure followed in HF clinics in the Copenhagen Region will fulfill the modified criteria for advanced HF from the HFA-ESC (primary end-point in the study)(Reference 1). Patients who are identified with advanced HF will be offered right heart catheterization, guided by ultrasound and inserted through the internal jugular vein, determining pulmonary capillary wedge pressure, cardiac index, central venous pressure, mean pulmonary artery pressure, and central venous oxygen saturation. Patients not fulfilling criteria for advanced HF will be offered right heart catheterization consecutively until 50 patients have been examined (this group will be a comparator group to the patients with advanced HF).

Patients identified with advanced HF will be offered listing for HTx or LVAD if an indication without a contraindication is present. Patients who fulfill the primary endpoint of modified HFA-ESC criteria for advanced HF, and are ineligible for, or unwilling to undergo HTx or LVAD implantation will be invited to participate in the SAINTS B study.

DETAILED DESCRIPTION:
Number of patients and sample size More than 3000 patients are followed in the HF clinics on Zealand including the greater Copenhagen region. The investigators plan to include 400 patients in the primary outcome analysis (SAINTS A) and hypothesize that 20% will fulfill the modified criteria for advanced HF.

Statistical analysis Descriptive statistics will be reported as mean +/- standard deviation (SD) or median (interquartile range (IQR)) depending on distribution. Comparisons between groups at baseline will be performed by unpaired t-tests for normally distributed continuous variables, by the Mann-Whitney U test (Wilcoxon rank-sum) for non-normally distributed continuous variables and χ2 or Fisher's exact test for categorical variables.

The primary outcome will be analyzed as the proportion n (%) of included patients who fulfill the modified HFA-ESC criteria for advanced HF. As for secondary outcomes, the investigators will analyze the proportion n (%) of patients who within the first 3 months are; 1) offered heart transplant listing, 2) offered LVAD implantation, 3) listed for HTx and 4) undergoing LVAD implantation. Further, comparisons of invasive hemodynamics, CPET measures, 6MWT, QoL and NTproBNP levels between patients with and without advanced HF will be made using an unpaired t-test or the Mann-Whitney U test for non-normally distributed continuous variables.

ELIGIBILITY:
Inclusion Criteria:

1. History of Chronic heart failure > 3 months
2. Stable (no hospitalization last 3 months) NYHA functional class II-III
3. HFrEF patients (Left ventricular ejection fraction (LVEF) ≤ 30%)
4. On or attempted betablocker and Renin-Angiotensin System (RAS) inhibitor treatment
5. Informed consent

Exclusion Criteria:

1. Body Mass Index (BMI) > 40 kg/m2
2. Chronic renal replacement therapy or estimated Glomerular Filtration Rate (eGFR) < 15 ml/min/1.73m2
3. Cardiac Resynchronization Therapy (CRT) implantation < 3 months ago or planned CRT
4. Severe primary valvular disease
5. On waiting list for heart transplantation or referred for evaluation
6. Cancer or other severe non-cardiac disease with estimated life expectancy less than 1 year

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed in Danish HF clinics in the Copenhagen region.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients screened who fulfill advanced HF criteria using a modified HFA-ESC definition | At time of screening
  Modified HFA-ESC criteria for advanced HF defined as:
  • LVEF ≤ 30% as estimated by echocardiography
  AND
  • Peak oxygen uptake (VO2peak) < 12 ml/kg/min (14 if on betablocker) with a Respiratory Exchange Ratio (RER) > 1.05 OR < 50% expected for age and gender OR 6 minute walk test (6MWT) distance < 300 meters
  AND
  • N-terminal pro B-type natriuretic peptide (NTproBNP) > 2000 pg / ml

SECONDARY OUTCOMES:
Proportion of patients offered heart transplant listing < 3 months after primary outcome | 3 months after meeting modified HFA-ESC criteria for advanced HF
Proportion of patients offered LVAD implantation < 3 months after primary outcome | 3 months after meeting modified HFA-ESC criteria for advanced HF
Proportion of patients listed for heart transplantation < 3 months after primary outcome | 3 months after meeting modified HFA-ESC criteria for advanced HF
Proportion of patients undergoing LVAD implantation < 3 months after primary outcome | 3 months after meeting modified HFA-ESC criteria for advanced HF
Pulmonary capillary wedge pressure (PCWP) in mmHg compared between patients with, and without advanced HF | Within 30 days from screening
  Measured during right heart catheterization
Cardiac index (CI) in l/min/m2 compared between patients with, and without advanced HF | Within 30 days from screening
  Measured during right heart catheterization
Central venous pressure (CVP) in mmHg compared between patients with, and without advanced HF | Within 30 days from screening
  Measured during right heart catheterization
Mean pulmonary artery pressure (mPAP) in mmHg compared between patients with, and without advanced HF | Within 30 days from screening
  Measured during right heart catheterization
Central venous oxygen saturation in % compared between patients with, and without advanced HF | Within 30 days from screening
  Measured during right heart catheterization
Peak oxygen uptake (VO2peak) in ml/kg/min compared between patients with, and without advanced HF | At time of screening
  Measured during cardiopulmonary exercise test
Peak respiratory exhange ratio compared between patients with, and without advanced HF | At time of screening
  The ratio between metabolic production of CO2 and the uptake of O2 measured during cardiopulmonary exercise test
Minute ventilation-to-carbon dioxide output slope (VE/VCO2) compared between patients with, and without advanced HF | At time of screening
  The ratio between metabolic production of CO2 and the uptake of O2 measured during cardiopulmonary exercise test
Peak Borg scale score compared between patients with, and without advanced HF | At time of screening
  The Borg scale score is a rating of perceived exertion on a scale from 6-20, with 6 representing at rest, and 20 the most strenuous exercise imaginable. Measured during cardiopulmonary exercise test
6 minute walk test compared between patients with, and without advanced HF | At screening
Quality of Life (Kansas City Cardiomyopathy Questionnaire (KCCQ) | At screening
NT-proBNP compared between patients with, and without advanced HF | At screening

CONTACTS AND LOCATIONS:
Overall Officials: Finn Gustafsson, MD, PhD, DMSci, Principal Investigator — Rigshospitalet, Denmark
Locations (6):
- Denmark (6):
  - Bispebjerg-Frederiksberg Hospital, Copenhagen
  - Amager/Hvidovre Hospital, Copenhagen
  - Herlev and Gentofte Hospital, Copenhagen
  - Glostrup Hospital, Glostrup Municipality
  - Nordsjællands Hospital Hillerød, Hillerød
  - Zeeland University Hospital Roskilde, Roskilde

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Crespo-Leiro MG, Metra M, Lund LH, Milicic D, Costanzo MR, Filippatos G, Gustafsson F, Tsui S, Barge-Caballero E, De Jonge N, Frigerio M, Hamdan R, Hasin T, Hulsmann M, Nalbantgil S, Potena L, Bauersachs J, Gkouziouta A, Ruhparwar A, Ristic AD, Straburzynska-Migaj E, McDonagh T, Seferovic P, Ruschitzka F. Advanced heart failure: a position statement of the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2018 Nov;20(11):1505-1535. doi: 10.1002/ejhf.1236. Epub 2018 Jul 17. PMID 29806100